CLINICAL TRIAL: NCT00814996
Title: Social Functioning in Schizophrenia
Status: Completed | Type: Observational
Sponsor: Far Eastern Memorial Hospital (Other)
Other Study IDs: FEMH-96-C-036
Record Dates: First submitted 2008-12-25; First posted 2008-12-29 (Estimated); Last update posted 2008-12-29 (Estimated); Status verified 2008-12

CONDITIONS: Schizophrenia
MeSH Terms: conditions — Schizophrenia

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective

GROUPS / COHORTS (2):
- 1: employment
- 2: unemployment

SUMMARY:
There are two research purposes of this study. One is to explore which psychosocial issue or biological issue would affect the social function among people with schizophrenia. The other one is to explore which social function would affect the job tenure among people with schizophrenia. There are 60 participants diagnosed with schizophrenia and divided into two groups, employment and unemployment. we will use several social function tests to collect social function, PANSS to evaluate their psychotic symptoms. And then we will compare and analysis the data through statistic software. Finally, we will have he answer about how social skills affect the social function and which social skill would affect the job tenure among people with schizophrenia.

ELIGIBILITY:
Inclusion Criteria:

* schizophrenia

Exclusion Criteria:

* substance abuse

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: schizophrenia
Sampling Method: Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2008-08; Primary Completion 2008-08 (Actual); Study Completion 2008-08 (Actual)